CLINICAL TRIAL: NCT06674824
Title: Role of Spectrophotometer in Early Prediction of Weaning Induced Cardiac Dysfunction
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Fouad, Assistant professor of anesthesia, intensive care and pain management, Ain Shams University
Other Study IDs: FMASU R238/2024
Record Dates: First submitted 2024-10-28; First posted 2024-11-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Weaning Failure
Keywords: Massimo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: massimo — measure plethysmography variability index in patients on spontaneous trial planning for extubation and evaluate its sensitivity in relation to transthoracic echocardiographic velocity time integral in early detecting weaning induced pulmonary edema

SUMMARY:
Weaning induced cardiac dysfunction is a common cause of weaning failure in critically ill patients. plethysmography variability index (PVI) is a non-invasive, real-time, and automated parameter for evalu¬ating fluid responsiveness.

By proving the validity of (PVI) in predicting successful spontaneous breathing trial Massimo can be used an easy noninvasive method that help in deciding the right time for weaning.

ELIGIBILITY:
Inclusion Criteria:

1. Intubation and mechanical ventilation
2. Fulfilling criteria for extubation
3. Fraction inspired oxygen less than 50%

Exclusion Criteria:

* a. Hemodynamic instability b. b. tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: intubated mechanically ventilated patients candidate for extubation
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
accuracy of change PVI in detecting volume responsiveness | 1 hour
  accuracy of change PVI in detecting volume responsiveness through measuring limits of agreement , Bias and correlation between PVI and a standard method of measurement which left ventricular outflow tract velocity time integral

SECONDARY OUTCOMES:
Sensitivity of trend of changes in hemoglobin by Massimo to detect WIPO and | 1 hour
time in minutes between rise of hemoglobin and clinical diagnosis of WIPO | 1 hour
  minutes between rise of blood hemoglobin concentration measured by Massimo and clinical diagnosis of WIPO

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt